CLINICAL TRIAL: NCT06895486
Title: A Phase 2, Randomized, Double- Dummy, Observer-Blind Study to Evaluate the Safety and Immunogenicity of Co-administered Novel Live Attenuated Monovalent Oral Poliomyelitis Vaccines in Healthy Young Infants Relative to Monovalent Vaccines Alone in Panama.
Brief Title: Study of Co-administered (Types 1 & 2) Novel Oral Poliomyelitis Vaccines Evaluation
Acronym: SCOPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); PT Bio Farma (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency); Technical Resources International, Inc. (TRI) (Unknown); Centro de Vacunación e Investigación (Cevaxin) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 109; U1111-1320-8206 (Registry Identifier: Universal Trial Number); RES-00751 (Other: PATH)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Poliomyelitis
Keywords: Vaccine; Polio; Poliomyelitis; novel oral polio vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Novel Oral Polio Vaccine Type 1 (nOPV1) and placebo (Experimental): nOPV1 and oral placebo (sterile water) given to 225 healthy infants
  Interventions: Biological: Novel Oral Polio Vaccine Type 1 (nOPV1); Biological: Placebo (Sterile Water)
- Group 2: Novel Oral Polio Vaccine Type 2 (nOPV2) and placebo (Experimental): nOPV2 and oral placebo (sterile water) given to 225 healthy infants
  Interventions: Biological: Novel Oral Polio Vaccine Type 2 (nOPV2); Biological: Placebo (Sterile Water)
- Group 3: nOPV1 and nOPV2 (Experimental): nOPV1 given along with nOPV2 to 225 healthy infants
  Interventions: Biological: Novel Oral Polio Vaccine Type 1 (nOPV1); Biological: Novel Oral Polio Vaccine Type 2 (nOPV2)

INTERVENTIONS:
Biological: Novel Oral Polio Vaccine Type 1 (nOPV1) — nOPV1 containing >10^7.0 CCID50 per dose
  Arms: Group 1: Novel Oral Polio Vaccine Type 1 (nOPV1) and placebo; Group 3: nOPV1 and nOPV2
Biological: Novel Oral Polio Vaccine Type 2 (nOPV2) — nOPV2 containing ≥10^5.0 CCID50 per dose
  Arms: Group 2: Novel Oral Polio Vaccine Type 2 (nOPV2) and placebo; Group 3: nOPV1 and nOPV2
Biological: Placebo (Sterile Water) — Sterile, nonpyrogenic preparation of water which contains no bacteriostat, antimicrobial agent, or added buffer
  Arms: Group 1: Novel Oral Polio Vaccine Type 1 (nOPV1) and placebo; Group 2: Novel Oral Polio Vaccine Type 2 (nOPV2) and placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of co-administration of nOPV1 + nOPV2 in infants, relative to those receiving monovalent nOPV vaccines alone and whether two and/or three doses of co-administered nOPV1 and nOPV2 are non-inferior to corresponding doses of nOPV1 alone and nOPV2 alone.

DETAILED DESCRIPTION:
This is a randomized, double dummy, observer blind, active comparator-controlled study. The study population will comprise healthy infants randomized at 16 weeks of age equally across three study groups, nOPV1 only group (N=225), nOPV2 only group (N=225) and co-administered nOPV1+ nOPV2 group (N=225). The participants in the nOPV1 and nOPV2 groups will receive concomitant oral placebo (sterile water) to blind the study arms for parents.

Participants will be screened (screening period 10 weeks), randomized and administered the first dose of study vaccine(s) at 16 weeks of age. The second and third dose of study vaccine(s) will be administered at 20 and 24 weeks of age, respectively. Participants will be consented and screened at 6 weeks of age and receive their routine Expanded Program on Immunization (EPI) vaccines by the study team. For each group, blood will be collected for immunologic testing at 16 (baseline), 20, 24, and 28 weeks of age. Serum specimens will be tested for humoral responses to vaccination by measurement of serum neutralizing antibody (NAb) according to established World Health Organization (WHO) protocols. Stool samples will be collected at various timepoints to evaluate type-specific shedding of polio virus following vaccination.

Following vaccination, participants will be monitored for at least 30 minutes for any immediate adverse events (AEs). Reactogenicity (solicited AEs) will be assessed during the 7 days (day of vaccination and 6 following days) after each vaccination. Parents will be given a post-immunization memory aid to record any local and systemic solicited reactions. In addition, data for unsolicited AEs will be collected for 28 days (day of study vaccination and 27 following days) after each vaccination. Data for SAEs will be collected throughout the study period following vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female infant 16 weeks (+ 7 days) of age, at the time of first study vaccination. Healthy as defined by the absence of any clinically significant medical condition or congenital anomaly as determined by medical history, physical examination, and clinical assessment by the investigator.
2. Parent(s) willing and able to provide written informed consent prior to performance of any study-specific procedure.
3. Resides in study area and parent understands and is able and willing to adhere to all study visits and procedures (as evidenced by a signed informed consent form (ICF) and assessment by the investigator).
4. Prior to study vaccination has received EPI vaccines as per the study EPI schedule and has received a single dose of IPV at 6 weeks (+7 days) of age.
5. Prior to study vaccination has received no doses of OPV, based upon no evidence of such vaccination per available documentation.
6. Parent agrees for participant to receive routine infant and childhood immunizations as per the approved protocol-adjusted schedule.

Exclusion Criteria:

1. Presence of anyone under 10 years of age in the participant's household (living in the same house or apartment unit) who does not have complete age appropriate vaccination status (as per local guidelines) with respect to poliovirus vaccines at the time of study vaccine administration.
2. Member of the participant's household (living in the same house or apartment unit) who has received OPV based on the vaccination records in the previous 3 months before study vaccine administration. Participants from household where a member received investigational nOPV3 vaccine will also be excluded from the study.
3. Low birth weight (LBW), defined as a birth weight of less than 2500 g (up to and including 2499 g) at the time of birth.
4. Premature birth (less than 37 weeks gestation).
5. From multiple births (due to increased risk of OPV transmissions between siblings).
6. Moderate or severe (grade ≥ 2) acute illness at the time of eligibility/first study vaccination - temporary exclusion. Note: Participants with mild (grade 1) acute illnesses may be considered eligible at the discretion of the investigator.
7. Presence of fever on the day of randomization/first study vaccination (axillary temperature ≥37.5˚C) - temporary exclusion.
8. Presence of abnormal vital signs (respiratory rate and/or heart rate) for age on the day of randomization/first study vaccination - temporary exclusion.
9. A known allergy, hypersensitivity, or intolerance to any components of the study vaccines, including all macrolide and aminoglycoside antibiotics (e.g., erythromycin and kanamycin).
10. Any reported known or suspected immunosuppressive or immunodeficiency condition (including HIV infection) in the participant or household member. Topical and inhaled steroids are permitted.
11. Receipt of any immune-modifying or immunosuppressant drugs prior to the first study vaccine dose or planned use during the study of study participants or a household member. Topical and inhaled steroids are permitted.
12. Any known or suspected bleeding disorder in the participant that would pose a risk to venipuncture or intramuscular injection.
13. Presence of severe malnutrition (weight-for- length/height z-score <-3SD median [per WHO published child growth standards]) - temporary exclusion if marginal and subsequently gains sufficient weight to attain z-score ≥-3 SD.
14. Receipt of any investigational product prior to the first administration of study vaccine, or planned use during the study period.
15. Receipt of rotavirus vaccine within 2 weeks prior to first study vaccination.
16. Prior receipt of an investigational product containing poliovirus vaccine.
17. Receipt of transfusion of any blood product or immunoglobulins prior to the first administration of study vaccine or planned use during the study period.
18. Parent or participant has any condition that in the opinion of the investigator would increase the participant's health risks in study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments).

Ages: 6 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 675 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious adverse events (SAEs) | From time of Dose 1 to end of study at Day 113
  Serious adverse event is any adverse event that results in any of the following outcomes: 1) Death, 2) Life-threatening, 3) Requires inpatient hospitalization or prolongation of existing hospitalization, 4) Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or 5) Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant or (and) require medical or surgical intervention to prevent one of the outcomes listed in the above
Frequency of solicited adverse events (AEs) | From time of vaccination until 7 days after Dose 1 (Day 8), Dose 2 (Day 36), and Dose 3 (Day 57)
  Solicited AEs are pre-specified AEs that are common or known to be associated with vaccination that are actively monitored as potential indicators of vaccine reactogenicity.
  The following solicited AEs will be monitored for this trial:
  Fever (axillary temperature ≥ 37.5°C), Vomiting, Diarrhea, Irritability or Abnormal Crying, Decreased feeding or appetite, and Fatigue or decreased activity
Frequency of unsolicited AEs | From time of vaccination to 28 days after Dose 1 (Day 29), Dose 2 (Day 57), and Dose 3 (Day 85)
  Unsolicited AEs are any AEs reported spontaneously by the participant's parent, observed by the study personnel during study visits or identified during review of medical records or source documents. In the absence of a diagnosis, abnormal physical examination findings or abnormal clinical safety laboratory test results that are assessed by the investigator to be clinically significant will be reported as an AE.
Percentage of participants demonstrating cumulative seroconversion of types 1 and 2 anti-polio serum neutralizing antibody (NAb) | 28 days after Dose 2 (Day 57)
  Cumulative Seroconversion is defined as type specific minimum 4-fold rise from baseline in those seropositive (NAb titer ≥1:8) at baseline, or post-vaccination seropositivity (titer ≥1:8) among those seronegative at baseline
Percentage of participants demonstrating cumulative seroconversion of types 1 and 2 anti-polio serum NAb | 28 days after Dose 3 (Day 85)
  Cumulative Seroconversion is defined as type specific minimum 4-fold rise from baseline in those seropositive (NAb titer ≥1:8) at baseline, or post-vaccination seropositivity (titer ≥1:8) among those seronegative at baseline

SECONDARY OUTCOMES:
Percentage of participants demonstrating cumulative seroconversion of type 1 and 2 anti-polio serum NAb | 28 days after Dose 1
  Cumulative Seroconversion is defined as type specific minimum 4-fold rise from baseline in those seropositive (NAb titer ≥1:8) at baseline, or post-vaccination seropositivity (titer ≥1:8) among those seronegative at baseline.
Median titer for type 1 and 2 anti-polio serum NAb | 28 days after Dose 1, Dose 2, and Dose 3
Geometric mean titer (GMT) for Types 1 and 2 anti-polio serum NAb | 28 days after Dose 1, Dose 2, and Dose 3
Post-vaccination GMT ratios of types 1 and 2 anti-polio serum NAb | Baseline compared to 28 days after Dose 1, Dose 2, and Dose 3
Type-specific and multitypic seroprotection*** rate. | 28 days after Dose 1, Dose 2, and Dose 3
  Seroprotection rate defined as anti-polio serum NAb reciprocal titer ≥ 8.
Geometric mean fold rise (GMFR) in NAb titer relative to baseline | Baseline compared to 28 days after Dose 1, Dose 2, and Dose 3
  For immunogenicity evaluation, baseline is defined as NAb measurement prior to the first nOPV dose at 16 weeks of age
GMFR in NAb titer following each dose relative to the pre-vaccination value. | Pre-vaccination titer compared to 28 days after Dose 1, Dose 2, and Dose 3
  For immunogenicity evaluation, baseline is defined as NAb measurement prior to the first nOPV dose at 16 weeks of age
Percentage of participants shedding types 1 and/or 2 polioviruses | At Day 1, Day 8, Day 29, Day 36, Day57, Day 64, Day 85 of the study
  Assessed by polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Saez Llorens, MD, Principal Investigator — Cevaxin
Locations (3):
- Panama (3):
  - Cevaxin - 24 de Diciembre, Panama City
  - Cevaxin - Ave. México, Panama City
  - Cevaxin - Chorrera, Panama City

IPD SHARING:
Plan to Share IPD: No